CLINICAL TRIAL: NCT05549323
Title: A PHASE 1B, TWO-PART, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER STUDY TO EVALUATE THE EFFICACY, SAFETY, AND PHARMACOKINETICS OF ORAL PF-07054894 IN ADULT PARTICIPANTS AGED 18-75 YEARS WITH MILD TO SEVERE ULCERATIVE COLITIS
Brief Title: A Study to Learn About the Safety, Effects and Pharmacokinetics of Study Medication (PF-07054894) for the Treatment of Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to business decision. The decision to terminate the trial was not based on any safety concerns associated with PF-07054894.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4151002; 2022-501047-32-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of the two groups in parallel for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group 1 (Experimental): Oral PF-07054894
  Interventions: Drug: PF-07054894
- Treatment Group 2 (Placebo Comparator): Matched Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07054894 — Oral
  Arms: Treatment Group 1
Drug: Placebo — Placebo
  Arms: Treatment Group 2

SUMMARY:
This is a study to learn if the experimental medicine (called PF-07054894) is safe, effective, and how it is processed in adult people with ulcers in the colon.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of moderate to severe (Part A) or mild to moderate (Part B) UC for ≥3 months prior to baseline.
* Active disease beyond the rectum (>15 cm of active disease from the anal verge at the screening endoscopy).

Part A (moderate to severe): Must have a 5 to 9 score on the modified mayo score, including an endoscopy subscore of at least 2. Part B (mild to moderate): Participants with mMS of 4 to 6, ES of ≥2 and RB score of ≥1

* Must have inadequate response to, loss of response to, or intolerance to at least one conventional therapy for UC.
* Total body weight >40 kg (88.2 lb).

Exclusion Criteria:

* Presence of indeterminate; microscopic; ischemic; infectious; radiation colitis; diverticular disease; Crohn's disease; colonic stricture; colonic obstruction/ resection; presence of cancer.
* History of bowel surgery within 6 months prior to baseline.
* History of significant trauma or major surgery within 4 weeks of screening or considered in imminent need of surgery or with elective surgery scheduled to occur during the study.
* Presence of clinical signs of fulminant colitis or toxic megacolon, primary sclerosing cholangitis and evidence of colonic dysplasia, adenomas or neoplasia.
* Clinically significant infections within 6 months of baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Part A: Proportion of participants achieving clinical remission at Week 12 in participants with moderate to severe UC. | Week 12
  Clinical remission based on modified Mayo Score is defined as endoscopic subscore equal 0 or 1 (without friability), stool frequency subscore equal 0 or 1, and rectal bleeding subscore equal 0
Part B: Percent change from baseline in the mMS in participants with mild to moderate UC. | Week 12

SECONDARY OUTCOMES:
Part A: Proportion of participants achieving improvement in endoscopic appearance at Week 12 | Week 12
  Endoscopic improvement is defined as a Mayo endoscopic subscore of ≤1 (without friability)
Part A: Proportion of participants with clinical remission at Week 12 | Week 12
  Clinical Remission defined by Total Mayo Score ≤2 and no individual subscore >1 and rectal bleeding subscore of 0
Part B: Proportion of participants achieving clinical remission at Week 12 | Week 12
  Clinical Remission based on modified Mayo Score is defined as endoscopic subscore 0 or 1 (without friability), stool frequency subscore 0 or 1, and rectal bleeding subscore 0.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (7):
  - IHS Health Research, Kissimmee, Florida
  - Kissimmee Endosocpy Center ( Endoscopy Only ), Kissimmee, Florida
  - Orlando Diagnostic Center ( CXR Only ), Kissimmee, Florida
  - Tampa Bay Endoscopy Center, Tampa, Florida
  - GCP Clinical Research, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Carta - Clinical Associates In Research Therapeutics Of America, San Antonio, Texas
- Germany (2):
  - Charité Research Organisation, Berlin
  - Charité Universitaetsmedizin Berlin - Campus Mitte, Berlin
- Poland (8):
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Medical Network Spółka z o.o. WIP Warsaw IBD Point Profesor Kierkuś, Warsaw, Masovian Voivodeship
  - KLIMED Marek Klimkiewicz, Bialystok, Podlaskie Voivodeship
  - MZ Badania Slowik Zymla Spolka Jawna, Knurów, Silesian Voivodeship
  - NZOZ Twoje Zdrowie EL Sp. z o. o., Elblag, Warmian-Masurian Voivodeship
  - Centrum Medyczne Med-Gastr, Lodz
  - IRMED, Piotrkow Trybunalski, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4151002